CLINICAL TRIAL: NCT00406692
Title: The Effects of Zonisamide on Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Clifford Knapp, PhD, Boston University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-25544
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Alcoholism
Keywords: Zonisamide; Alcoholism; Alcohol
MeSH Terms: conditions — Alcoholism | interventions — Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zonisamide (Experimental): In open-label non-placebo controlled trial subjects are treatment with zonisamide 400 mg during the maintenance phase of this study
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — Week 1 (Wk1) -100 mg daily; Wk 2- 100 mg daily; Wk 3- 200 mg daily; Wk 4- 200 mg daily; Wk 5- 300 mg daily; Wk 6- 300 mg daily; Wk 7-11- 400 mg daily; Wk 12(Days 1-5) 300 mg daily; Wk 12 (Day 6-7) Week 13 (Days 1-3)- 200 mg daily; Week 13 (Days 4-7) - 100 mg daily.

SUMMARY:
In this study the influence of zonisamide administration over a 13 week period on alcohol consumption in alcoholic (alcohol dependent) subjects will be examined. The dose of zonisamide given to subjects will be slowly increased over a period of several weeks. They will receive a full dose over a 5 week period. This will be a pilot study in which all of the subjects will only receive zonisamide. A primary objective of this study is to determine the possible size of the effect that zonisamide administration has on drinking (i.e. drinks consumed per day) to allow us to plan for a larger clinical trial of the effects of zonisamide on alcohol dependence.

ELIGIBILITY:
INCLUSION CRITERIA

To be admitted into this study patients must meet the following criteria:

1. DSM IV TR Diagnosis of Alcohol Dependence; minimal level of 14 drinks per week for women or 21 drinks per week for men over a 28 day consecutive period during the 90 day period prior to the screening session.
2. Male or Female 21-64 years of age.
3. Able to provide informed consent and comprehend study procedures.
4. Negative urine toxicological screen for opioids, psychomotor stimulants, sedative-hypnotics, and cannabinoids. If the urine tox screen was positive for any substance it may be repeated within two weeks.
5. Score of >8 on the Alcohol Use Disorder Identification Test (AUDIT) during screening.
6. Must be suitable for outpatient management of alcoholism.
7. Express desire to stop drinking or reduce alcohol consumption with a possible long-term goal of abstinence.
8. Provide contact information for themselves or an alternate contact that the staff will call in case of missed appointment.
9. Women must be postmenopausal for at least one year, be surgically sterile, be using an effective method of birth control (e.g. contraceptive injection, intrauterine device, spermicide with barrier, contraceptive patch, contraceptive ring, male partner sterilization, oral contraceptives) or completely abstinent (and agree to use one of the above mentioned methods of contraception if sexual activity is ever initiated).
10. Must be able to take oral medications, adhere to the regimen and be willing to return for follow up visits.
11. Must have breath alcohol concentration of no more than 0.01% when the informed consent is provided and the consent form is signed.
12. Must have resided at the same address for at least 3 months.

EXCLUSION CRITERIA

Patients meeting the following criteria will be excluded from the study:

1. Dependent on or extensive abuse of drugs or substances other than ethanol, nicotine, or caffeine.
2. DSM IV-TR diagnosis of any current Axis I diagnosis other than alcohol dependence, nicotine dependence, or caffeine dependence that in the opinion of the study physicians might require intervention with either pharmacological or non-pharmacological therapy that will interfere with the course of the study.
3. Receiving inpatient or outpatient treatment for alcohol dependence (with the exception of AA or other self-help groups) within 4 weeks prior to enrollment into this study.
4. Subjects with a score of 10 or greater on the CIWA-Ar (a withdrawal scale) on first or second visits.
5. Currently being treated with acamprosate, disulfiram or naltrexone.
6. Currently being treated with any of the following medications: a) Antipsychotic agents- including clozapine, risperidone, quetiapine, haloperidol b) Antimanic or anticonvulsant agents- including lithium carbonate, phenytoin, phenobarbital, carbamazepine, topiramate, valproic acid, divalproex, tiagabine c) Sedative-hypnotic or antianxiety agents-including triazolam, temazepam, zolpidem, zalepron, buspirone, alprazolam, diazepam, clonazepam, oxazepam, lorazepam d) chronic opioid treatment- including methadone, buprenorphine, oxycodone, morphine e) Psychomotor stimulants- amphetamine derivatives, methylphenidate
7. Subjects who are legally mandated to participate in an alcohol treatment program
8. Use of any medication known to inhibit or induce cytochrome P450 3A4 enzymes including macrolide antibiotics, fluoxetine, and carbamazepine.
9. Subjects who have attempted suicide or who have had suicidal ideation within 30 days of their first visit as assessed using responses from the SCID and Hamilton Depression scale.
10. Subjects with renal disease (including severe infection and cancer), impaired renal clearance (CrCl less than 50 ml/min), or history of kidney stones.
11. Subjects with AST or ALT >3 times the upper limit of the normal range during screening.
12. History of significant neurological disorder, including a history of seizures, stroke, dementia, multiple sclerosis, Parkinson's disease, brain tumors, or encephalitis.
13. Subjects who are pregnant (as assessed by serum HCG) or lactating.
14. Subjects known to have clinically significant medical conditions. These may include: symptomatic CAD or PVD, malignancy or history of malignancy in the last 5 years, significant pulmonary disease or endocrinological disorders.
15. Subjects with prior hypersensitivity to zonisamide or related compounds, including sulfonamides (e.g. sulfisoxazole) carbonic anhydrase inhibitors (e.g. acetazolamide), sulfonylureas (e.g. chlorpropamide), sulfamates (e.g. topiramate), thiazide (e.g. hydrochlorothiazide), and loop diuretics (e.g. furosemide) except ethacrycrynic acid.
16. Subjects who in the opinion of the study physicians should not be enrolled based on the precautions, warnings, and contraindications stated on the package insert for zonisamide.
17. Impending incarceration.
18. Score of 25 or less on the Folstein Mini-Mental examination.
19. History of anticonvulsant-induced rash.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Knapp, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was from May 2007 to April 2008. The primary forms of recruitment were newspaper advertisement and radio advertisement.
Groups:
- Zonisamide: 400 mg daily
Period: Overall Study
Arm/Group | Zonisamide
Started | 16
Completed | 9
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zonisamide
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: The Weekly Mean Number of Standard Drinks Consumed Per Day at Baseline and Treatment Phase
Description: The mean daily standard alcoholic drinks were determined for the baseline period and each treatment week as a measure of alcohol intake. One standard drink=14g of alcohol. Mean value is the difference between mean standard drinks for the baseline period and week 12 of the study.
Time Frame: Baseline and Week 12
Population: ITT
Measure: Mean (Standard Error); unit: Standard Drinks
Arm/Group | Zonisamide
Number analyzed (Participants) | 16
Standard Drinks | -6.7 (1.5)
Statistical Analysis 1: Comparison: Zonisamide; Null Hypothesis: No difference in the mean daily standard drinks consumed between the baseline period and the zonisamide treatment weeks; Test type: Superiority or Other; p < 0.0003, Mixed Models Analysis — Null Hypothesis: No difference in the mean daily standard drinks consumed for the baseline period and the zonisamide treatment weeks; Mean Difference (Final Values) = -6.7, Standard Error of Mean 1.5

2. Primary Outcome: Difference in Mean Words for the Phonetic Portion of the Controlled Word Association Test (COWAT).
Description: Subjects were asked to generate as many words as possible starting with a particular letter over a 60 second period. Three letters were used for each sessions. Values shown are the differences between values obtained for the baseline and week 12 test session.
Time Frame: Week 0- Baseline and Week 12
Population: ITT
Measure: Mean (Standard Error); unit: Number of Words
Arm/Group | Zonisamide
Number analyzed (Participants) | 16
Number of Words | -6.4 (3.9)
Statistical Analysis 1: Comparison: Zonisamide; Null Hypothesis: No significant change in the mean number of words produced during phonetic portion of the Controlled Word Association Test between the baseline period and the treatment weeks; Test type: Superiority or Other; p < 0.22, Mixed Models Analysis; Mean Difference (Net) = -6.7, Standard Error of Mean 3.9

3. Secondary Outcome: Symbol Digit Modalities Test (DSMT)
Description: Number of correct digit substitutions on the DSMT per session with the possible maximum score being 188. The value shown is for difference between mean scores obtained for baseline and week 12 sessions.
Time Frame: Baseline, Week 12
Population: ITT
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Zonisamide
Number analyzed (Participants) | 16
Units on a scale | -1.5 (4)
Statistical Analysis 1: Comparison: Zonisamide; Null Hypothesis: No significant difference for mean scores obtained for baseline, week 4 and week 12; Test type: Superiority or Other; p < 0.55, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, Standard Error of Mean 4

ADVERSE EVENTS:
Time Frame: 13 Weeks
Arm/Group | Zonisamide
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=16)
Sedation (Nervous system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Limitations of this trial include lack of a placebo controlled arm and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes